CLINICAL TRIAL: NCT05340985
Title: Investigating the Effects of Hydroxyvitamin D3 Versus Vitamin D3 on Clinical, and Radiologic Progress and Th17/Tregs Balance in MS Patients: A Randomized, Clinical Trial- a Pilot Study
Brief Title: Investigating the Effects of Hydroxyvitamin D3 on Multiple Sclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1400-3-233-56129
Record Dates: First submitted 2022-03-02; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Adult ALL; Vitamin D3 Deficiency
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Calcifediol; Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial with a parallel group and allocation 1:1.
Who Masked: Outcomes Assessor
Masking Description: All participants at the MS clinic will be blinded to trial intervention allocation. The main outcomes will be evaluated by neurologists.
  Investigator is also blind; two type of vitamin D; 25(OH)D3 and cholecalciferol capsules with similar shape and color.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 25(OH)D3 (Calcifediol) (Experimental): 50 micrograms per day 25(OH)D3 or vitamin D hydroxylated for 24 weeks
  Interventions: Dietary Supplement: 25(OH)D3
- Cholecalciferol (Experimental): 50 micrograms (2000IU) per day Cholecalciferol for 24 Weeks
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: 25(OH)D3 — calcifediol
  Other Names: vitamin D analog
  Arms: 25(OH)D3 (Calcifediol)
Dietary Supplement: vitamin D3 — Cholecalciferol
  Other Names: activated 7-dehydrocholesterol
  Arms: Cholecalciferol

SUMMARY:
Investigating the effects of hydroxyvitamin D3 on clinical, radiologic and immunomodulatory markers in MS patients: A randomized, clinical trial- a pilot study

DETAILED DESCRIPTION:
Vitamin D deficiency/insufficiency is a risk factor for developing MS and is linked to increased disease activity in those with established disease. Several clinical trials have already been conducted to consider the effect of vitamin D supplementation on clinical outcomes of the disease but the findings were inconsistent.

This paradox may be explained by supplementation dose, trial duration and also an insufficient rise in serum 25-hydroxyvitamin D to be effective on immunomodulatory pathways and consequent clinical outcomes.

Of note, it was revealed that MS patients have a lower rise in serum 25-hydroxyvitamin D [25(OH)D] levels compared with healthy controls (HCs), when given the same amount of oral cholecalciferol supplementation.

Cholecalciferol is the main vitamin D supplement that was used in these trials. When vitamin D3 is ingested, it is incorporated into chylomicrons and enters the lymphatic system. The chylomicrons then enter into the bloodstream via the superior cava. Most of the vitamin D is incorporated into the body fat.

Vitamin D3 in the circulation and the vitamin D3 that is slowly released from the body fat into the circulation is converted in the liver to 25(OH)D3, taking approximately 6-8 weeks to achieve a steady state concentration of 25(OH)D3.

The more rapid increase in serum concentrations of 25(OH)D3, by treatment with calcifediol instead of cholecalciferol, may provide an advantage through rapid entry into its target innate and adaptive immune cells, resulting in the paracrine/autocrine production of 1α,25(OH)2D which interacts with the vitamin D receptor (VDR) to modulate immune function.

ELIGIBILITY:
Inclusion Criteria:

1. MS type: relapsing-remitting MS (RRMS)
2. older than 18 year-old
3. Vitamin D deficiency/insufficiency (25(OH)D<30 ng/ml

Exclusion Criteria:

1. medications or disorders that would affect vitamin D metabolism
2. history of other chronic disorders
3. history of conditions that could lead to high serum calcium levels
4. pulse therapy in the last 3 months
5. history of attack in the last 3 months
6. using corticosteroid in the last 3 months
7. be pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on ID
Enrollment: 54 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of relapses | 6 months (baseline and end of 6th month) in each intervention arm
  neurologic symptoms lasting more than 24 hours which occur at least 30 days after the onset of a preceding event
disability | 6 months (baseline and end of 6th month) in each intervention arm
  Change in expanded disability status scale (EDSS) according to Kurtzke 1983. The minimum is 0 (no disability) and maximum value is 10 (Death due to MS)- higher scores mean a worse outcome.
Change in MRI parameters | 6 months (baseline and end of 6th month) in each intervention arm
  new lesions on T2 weighted images, gadolinium enhancing lesions in T1-weighted images
changing in brain parameters of Diffusion tensor imaging (DTI) | 6 months (baseline and end of 6th month) in each intervention arm
  the integrity of white matter (WM) by analyzing WM microstructure through DTI
changing in Cognition | 6 months (baseline and end of 6th month) in each intervention arm
  Changing in cognitive functions by the Minimal Assessment of Cognitive Function in MS (MACFIMS) battery. The lower the score the more disfunction.
  MACFIMS is consisting of 7 subtests including:
  1. the California Verbal Learning Test second edition (CVLT-II), with the range score: 0-80
  2. the Paced Auditory Serial Addition Test (PASAT), with the range score: 0-16
  3. the Symbol Digit Modalities Test (SDMT), with the range score: 0-110
  4. the Brief Visuospatial Memory Test-Revised (BVMT-R), with the range score: 0-36
  5. the Controlled Oral Word Association Test (COWAT), with the range score: 0-12
  6. the Delis-Kaplan Executive Function System (DKEFS) sorting Test, with the range score: 0- undetermined
  7. the Judgment of Line Orientation Test (JLO), with the range score: 0-30
  The higher score in each subtest means the better cognitive function
CD4+ T cell response | 6 months (baseline and end of 6th month) in each intervention arm
  After six months, changing the balance of Th17 and Tregs subtypes of CD4+ T cells.
  Detecting interleukin (IL) 17 -expressing T cells and Tregs expressing T cells by flow cytometry.
Differential gene expression | 6 months (baseline and end of 6th month) in each intervention arm
  After six months of 25-hydroxy vitamin D supplementation, the differentially expressed genes (DEGs) in peripheral blood mononuclear cells at the transcriptome level will be considered by RNA-seq

SECONDARY OUTCOMES:
needing hospitalization | 6 months (baseline and end of 6th month) in each intervention arm
  needing hospitalization due to remissions and exacerbations of the disease
changing in quality of life | 6 months (baseline and end of 6th month) in each intervention arm
  changing in quality of life that determined by the Short Form Health Survey that contains 36-item (Sf36). The score is between 0-100.
  The lower the score the more disability. The higher the score the less disability.
effective in rapidly raising circulating levels of 25(OH)D3 | 6 months (baseline and end of 6th month) in each intervention arm
  Serum levels of 25-hydroxy vitamin D (25(OH)D will be measured by High-performance liquid chromatography (HPLC)
changing in the circulating levels of interleukin 17 as a inflammatory marker | 6 months (baseline and end of 6th month) in each intervention arm
  After six months of calcifediol/or cholecalciferol supplementation, measuring serum levels of IL-17 by enzyme-linked immunoassay (ELIZA) kit.
changing in the levels of interleukin 10 as anti- inflammatory marker | 6 months (baseline and end of 6th month) in each intervention arm
  After six months of calcifediol/or cholecalciferol supplementation, measuring serum levels of IL-10 by ELIZA kit.
changing in the levels of Tumor Necrosis Factor alpha (TNF-a) as an inflammatory marker related the T-CD4 subsets | 6 months (baseline and end of 6th month) in each intervention arm
  After six months of calcifediol/or cholecalciferol supplementation, measuring serum levels of TNF-a by ELIZA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamadali Sahraian, MD, Study Chair — Multiple Sclerosis Research Center, Tehran University of Medical Sciences; Zhila Maghbooli, PhD, Principal Investigator — Multiple Sclerosis Research Center, Tehran University of Medical Sciences; Michael F Holick, PhD,MD, Principal Investigator — Boston University